CLINICAL TRIAL: NCT01863290
Title: Transitions Clinic Network: Linking High-Risk Medicaid Patients From Prison to Community Primary Care
Brief Title: Linking Former Inmates to Primary Care
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1301011280
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Hypertension; Substance Abuse; Asthma; Depression
Keywords: prison; reentry; health care utilization
MeSH Terms: conditions — Hypertension; Substance-Related Disorders; Asthma; Depression; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Former inmates: Former inmates with a chronic disease condition or aged 50 years and above engaged into primary care through an innovative primary care redesign model of the Transitions Clinic Network.
  Interventions: Other: Primary care redesign

INTERVENTIONS:
Other: Primary care redesign — Connect individuals released from prison to primary care using trained, culturally competent primary care providers and community health workers (CHWs).

SUMMARY:
The Transitions Clinic Network (TCN)aims to connect former inmates to primary care using trained, culturally competent primary care providers and community health workers (CHWs). The purpose of this project is to support ongoing quality improvement at the 13 participating sites by training culturally competent CHWs and measuring the health, health care utilization, and the costs of caring for former inmates.

DETAILED DESCRIPTION:
The Transitions Clinic Network (TCN) is a network of 13 community-based transitional healthcare programs, which aim to improve health, improve health care, and lower costs for vulnerable, high-risk Medicaid patients returning from prison across the United States. The TCN aims to connect individuals released from prison to primary care using trained, culturally competent primary care providers and community health workers (CHWs). The providers and CHWs, help patients obtain timely healthcare; promote healthy reintegration into their communities; provide care coordination and chronic disease management; and prevent unnecessary emergency department utilization and hospitalizations.

The project supports ongoing quality improvement at each of the 13 clinical sites by measuring the health, health care utilization, and the costs of caring for recently released patients. We will prospectively examine the rates of primary care engagement, acute care utilization, substance abuse and reported health, and recidivism in a cohort of 2000 patients recently released from prison receiving primary care at the 13 TCN programs. We will compare these rates of utilization at 6, 12, 18, 24, 30, 36 months to patient self-reported utilization prior to incarceration and historical controls.

Additionally, we aim to describe the implementation of, fidelity to, and sustainability of the TCN model in each of these clinical programs. Specifically, we aim to capture assets and barriers to starting and sustaining primary care programs targeting returning prisoners.

ELIGIBILITY:
Inclusion Criteria:

* Recently-released from prison (within one month)
* Has >=1 chronic disease condition , and/or age >=50 years
* Plans to live in the TCN area for the duration of the study
* Understands English or Spanish and able to provide consent

Exclusion Criteria:

* Does not plan to live in the TCN area for the duration of the study
* Does not understand English or Spanish, or unable to provide consent
* Does not plan to receive healthcare through a TCN clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Former inmates; released from state or federal prisons.
Sampling Method: Non-Probability Sample
Enrollment: 816 (Actual)
Dates: Start 2013-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Health outcomes | One year
  Patient health outcomes and quality of life, including self reported health, depression severity, hypertension, and relapse to alcohol and substance use.

SECONDARY OUTCOMES:
Cost savings to the Centers for Medicare & Medicaid Services | 3 years
  Cost savings from prevented emergency department visits and hospitalizations, as well as improved health and decreased recidivism
Health care utilization | One year
  Rates of engagement with primary care, all cause emergency department utilization and hospitalization rates, emergency department utilization and hospitalization rates for ambulatory care sensitive conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Emily A Wang, MD, MAS, Principal Investigator — Yale University
Locations (11):
- United States (10):
  - University of Alabama, Birmingham, Alabama
  - Contra Costa Health Services (East and West Contra Costa), Martinez, California
  - Southeast Health Center, San Francisco, California
  - Santa Clara Health Center, San Jose, California
  - Yale Primary Care Center, New Haven, Connecticut
  - East Baltimore Medical Center, Baltimore, Maryland
  - Boston Healthcare for the Homeless Program, Boston, Massachusetts
  - Morningside Clinic, New York, New York
  - Montefiore Transition Clinic, New York, New York
  - Medicine in Psychiatry Service clinic of the University of Rochester Medical Center, Rochester, New York
- Corporacion SANOS, Caguas, Puerto Rico

REFERENCES:
- [Derived] Redmond N, Aminawung JA, Morse DS, Zaller N, Shavit S, Wang EA. Perceived Discrimination Based on Criminal Record in Healthcare Settings and Self-Reported Health Status among Formerly Incarcerated Individuals. J Urban Health. 2020 Feb;97(1):105-111. doi: 10.1007/s11524-019-00382-0. PMID 31628588